CLINICAL TRIAL: NCT03872934
Title: Effect of Different Music Types on Implant Surgery Anxiety - Randomized Controlled Study
Brief Title: Effect of Different Music Types on Implant Surgery Anxiety
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Erzincan University (Other)
Responsible Party: Principal Investigator, ILKE KUPELI, assist. prof., Erzincan University
Other Study IDs: EBYU 1
Record Dates: First submitted 2019-03-08; First posted 2019-03-13 (Actual); Last update posted 2019-07-15 (Actual); Status verified 2019-07

CONDITIONS: Anxiety, Dental
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Turkish music group: Turkish music group (Saba or rast makam)
  Interventions: Behavioral: implant anxiety
- classical western music: classical western music (vivaldi)
  Interventions: Behavioral: implant anxiety
- soft rock music: soft rock music (elvis)
  Interventions: Behavioral: implant anxiety
- control group (group not listening music): control
  Interventions: Behavioral: implant anxiety

INTERVENTIONS:
Behavioral: implant anxiety — to determine the type of music that reduces anxiety in patients undergoing implant surgery.

SUMMARY:
A general term, dental anxiety, is defined as fear or an abnormal concern to visit the dentist for unwanted concerns about preventive care and dental procedures. anxiety; dental examinations or treatment can be prevented or postponed.

This delay in dentistry typically leads to much more serious dental problems, often leading to more expensive, more invasive and possibly emergency treatment. Therefore, reducing anxiety is important both in terms of patient, physician and cost.

ELIGIBILITY:
Inclusion Criteria:

* Will undergo elective implant surgery,
* between 40-70 years

Exclusion Criteria:

* Who does not agree to participate in the study,
* Under 40, over 70 years,
* Patients with ear disorders (ie, not suitable for musical intervention),
* arrhythmia
* patients with physical condition III or higher (American Society of Anesthesiologists)

Ages: 40 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Eighty patients aged 40-70 years will undergo elective implant surgery.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2019-07-15 (Estimated); Primary Completion 2019-12-15 (Estimated); Study Completion 2020-01-15 (Estimated)

PRIMARY OUTCOMES:
Corah's dental anxiety scale | six month
  the type of music that reduces anxiety in patients undergoing implant surgery.

CONTACTS AND LOCATIONS:
Overall Officials: ilke kupeli, Principal Investigator — Erzincan University

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Miyata K, Odanaka H, Nitta Y, Shimoji S, Kanehira T, Kawanami M, Fujisawa T. Music before Dental Surgery Suppresses Sympathetic Activity Derived from Preoperative Anxiety: A Randomized Controlled Trial. JDR Clin Trans Res. 2016 Jul;1(2):153-162. doi: 10.1177/2380084416650613. PMID 30931796
- [Result] Bodner E, Iancu I. Recalling the threat: dental anxiety in patients waiting for dental surgery. Isr J Psychiatry Relat Sci. 2013;50(1):61-6. PMID 24029113
- [Result] Thoma MV, Zemp M, Kreienbuhl L, Hofer D, Schmidlin PR, Attin T, Ehlert U, Nater UM. Effects of Music Listening on Pre-treatment Anxiety and Stress Levels in a Dental Hygiene Recall Population. Int J Behav Med. 2015 Aug;22(4):498-505. doi: 10.1007/s12529-014-9439-x. PMID 25200448
- [Result] Wright H. The Correlation of Classical, Jazz, and Pop Music to a Reduction of Dental Anxiety Experienced by Adult Patients. 2018.
- See also: Encyclopedia of Medical Concepts. Reference. MD website. — http://www.reference.md/files/D016/mD016854.html